CLINICAL TRIAL: NCT03108976
Title: Build-up of Action Representation During Neurodevelopment: Dysfunctions in Autism Spectrum Disorders?
Brief Title: Build-up of Action Representation in Autism Spectrum Disorders
Acronym: ASD-BARN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL16_0677
Record Dates: First submitted 2017-03-30; First posted 2017-04-11 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Healthy; Autism Spectrum Disorder
Keywords: Autism; Sensori-motor learning; Development; Neuroimaging
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Magnetoencephalography; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): Children with a typical development.
  Interventions: Other: Behavioral assessments; Other: Magnetoencephalography (MEG); Other: Magnetic Resonance Imaging (MRI)
- Case group (Active Comparator): Children with Autism Spectrum Disorders.
  Interventions: Other: Behavioral assessments; Other: Magnetoencephalography (MEG); Other: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Other: Behavioral assessments — Kinematics measures, concomitant to Magnetoencephalography (MEG, measures oscillatory rhythms in the brain) and Magnetic Resonance Imaging (MRI, used to provide an anatomical image of each participant's brain to be coregistered with oscillatory measurements) recordings, enable to track sensori-motor learning based on performance, and oscillatory changes (with high temporal and spatial resolution).
Other: Magnetoencephalography (MEG) — Kinematics measures, concomitant to Magnetoencephalography (MEG, measures oscillatory rhythms in the brain) and Magnetic Resonance Imaging (MRI, used to provide an anatomical image of each participant's brain to be coregistered with oscillatory measurements) recordings, enable to track sensori-motor learning based on performance, and oscillatory changes (with high temporal and spatial resolution).
Other: Magnetic Resonance Imaging (MRI) — Kinematics measures, concomitant to Magnetoencephalography (MEG, measures oscillatory rhythms in the brain) and Magnetic Resonance Imaging (MRI, used to provide an anatomical image of each participant's brain to be coregistered with oscillatory measurements) recordings, enable to track sensori-motor learning based on performance, and oscillatory changes (with high temporal and spatial resolution).

SUMMARY:
Autistic spectrum disorders (ASD) are highly debilitating developmental syndromes which core feature is social and communications disorders. Motor skill impairments are frequently described in autism, but few studies have addressed the question of their origin and their specificity. Furthermore, it is not clear whether motor problems encountered in autism are related to dyspraxia, or if they present with specific features. This project aims at deciphering the origin of motor problems encountered by children who grow-up with autism in order to propose early interventions that could influence the other developmental trajectories, such as the social one.

Brain dynamics during sensori-motor learning is explored by applying magnetoencephalography (MEG) during the Bimanual Load-Lifting paradigm. Different motor processes namely: proprioceptive monitoring, use and update of a sensori-motor representation, anticipatory executive control will be correlated to brain oscillation modulation, both topographically and temporally. Two groups of children (aged between 7 and 12) are compared: a group of children with ASD and a control group of typically developing children.

ELIGIBILITY:
Inclusion Criteria:

* Control group: children aged between 7 and 12
* Case group: children aged between 7 and 12 with a diagnostic of Autism Spectrum Disorders

Exclusion Criteria:

* Control group: presence of a neurological pathology, mental retardation or language and motor developmental delay
* Case group: presence of a neurological pathology, mental retardation

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2015-04-10 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Changes of cerebral oscillations in three frequency bands (alpha, beta, gamma) during sensori-motor learning. | Day 1
  Oscillatory measures are computed in the sensor and source space in order to identify the regions involved in the sensori-motor learning in the control group and in the ASD group.

SECONDARY OUTCOMES:
Correlation between oscillatory measures and learning performance. | Day 1
  Kinematic recordings enable to measure the learning performance at the end of the experiment. This measure will be correlated with oscillatory changes during the task.

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine SONIE, MD, Principal Investigator — CH le Vinatier
Locations (1):
- CH le Vinatier, Bron, France